# DBT Skills Training for Adults with Autism Spectrum Disorder and Emotion Regulation Difficulties

30.01.2025

## **Request for Participation in Research Project**

DBT SKILLS TRAINING FOR ADULTS WITH AUTISM SPECTRUM DISORDER AND DIFFICULTIES in EMOTION REGULATION

#### PURPOSE OF THE PROJECT AND WHY YOU ARE BEING ASKED

An increasing number of adults are discovering that they have Autism Spectrum Disorder (ASD). Despite the growing number of adults with ASD, there is a significant lack of treatment options for them. Difficulties with emotion regulation are increasingly recognized as central challenges for many adults with ASD. Difficulties in Emotion regulation can include the inability to recognize, understand, and manage emotions, which may lead to behaviors that negatively influence your life. These may include difficulties regulating impulses, engaging in: self-harm, aggressive behavior, violence, and avoidance. Developing effective strategies to manage difficult emotions can improve the quality of life for people with ASD.

DBT skills training is designed to help individuals who struggle with intense emotions and destructive behaviors. DBT skills training has proven effective for various disorders and has shown positive effects in reducing self-harm among adults with ASD. The goal of the skills training is to learn how to manage intense emotions, difficult relationships, and crises to more easily achieve life goals.

You are being offered participation because you have ASD and are receiving treatment at the Psychiatric Outpatient Clinic in Molde.

## WHAT DOES THE PROJECT INVOLVE?

Participation in this project involves attending weekly DBT skills training sessions over a 6-month period (26 sessions). The training takes place in a group of 4–6 participants, each session lasting two hours. You will learn practical skills to help manage difficult emotions, increase mindfulness, reduce stress levels, and maintain relationships with others. This offer is in addition to your regular treatment with your primary therapist.

You will be asked to complete weekly skills tracking sheets and fill out questionnaires at the beginning and end of the training. The purpose is to assess your experience with the program, its relevance, feasibility, and whether you benefited from the treatment. As part of this, you will be asked questions about destructive behavior, difficulties managing emotions, and your personal experiences. We will also collect diagnostic and demographic

information (age, living situation, marital status, childcare responsibilities, employment status).

The project will collect and register information about you. We will use interviews and questionnaires, along with diagnostic information from your medical records. This information will be used to develop a new treatment offering for adults with ASD.

#### **POSSIBLE BENEFITS AND RISKS**

Participants in the project are likely to develop better skills for managing difficult emotions without resorting to destructive behavior. Weekly group attendance and practicing new skills may be demanding but also rewarding if successful. Participation may lead to improved services for adults with ASD and emotion regulation difficulties. It may help us improve treatment offerings for you and others with similar challenges within the Mental Health Clinic at Helse Møre og Romsdal.

## **VOLUNTARY PARTICIPATION AND WITHDRAWAL OF CONSENT**

Participation in the project is voluntary. If you wish to participate, you must sign the consent form on the last page. You may withdraw your consent at any time without giving a reason. This will not affect your continued treatment. If you withdraw, you may request that your collected data be deleted, unless it has already been included in analyses or used in scientific publications.

If you later wish to withdraw or have questions about the project, you may contact:

- Johanna Vigfusdottir, Clinical Psychologist, DBT Team Email: johanna.vigfusdottir@helse-mr.no | Phone: 467 46 154
- Reidun Høidal, Clinical Psychologist, DBT Team Email: reidun.hoidal@helse-mr.no | Phone: 917 80 504
- Project Leader: Egil Jonsbu, Chief Physician

Email: egil.jonsbu@helse-mr.no

#### WHAT HAPPENS TO YOUR INFORMATION?

The information collected about you will only be used as described in the project's purpose. You have the right to access the information registered about you and to correct any errors. You also have the right to know about the security measures in place for handling your data.

All data will be processed without names, personal ID numbers, or other directly identifying information. A list linking names to participant numbers is the only connection between your data and your identity. Only psychologists Reidun Høidal and Johanna Vigfusdottir have access to this list.

The project is planned to conclude in 2027. After the research ends, your data will be stored for five years for control purposes. Any extension of use or storage time requires approval

from REK and other relevant authorities. You may file a complaint about the handling of your data with the Data Protection Authority or the institution's Data Protection Officer.

## **FOLLOW-UP PROJECT**

If a follow-up project becomes relevant, you may be contacted again after the treatment ends.

If you need to talk to someone as a result of participating in the project, you may contact:

- Reidun Høidal, Clinical Psychologist | Phone: 917 80 504
- Johanna Vigfusdottir, Clinical Psychologist | Phone: 467 46 154

#### **INSURANCE**

The Patient Injury Act applies as usual.

#### **APPROVAL**

The Regional Committee for Medical and Health Research Ethics has reviewed and preapproved the project (#836937).

Helse Møre og Romsdal and Project Leader Chief Physician Egil Jonsbu are responsible for data protection in the project.

We process your data based on your consent. You have the right to complain to the Data Protection Authority.

#### **CONTACT INFORMATION**

If you have questions about the project, you may contact:

- Johanna Vigfusdottir, Clinical Psychologist, DBT Team: johanna.vigfusdottir@helse-mr.no
- Reidun Høidal, Clinical Psychologist, DBT Team: reidun.hoidal@helse-mr.no
- Section Leader: Tonje Sæter: tonje.seter@helse-mr.no
- Data Protection Officer: Jan Rino Austdal: jan.rino.austdal@helse-mr.no

#### **CONSENT**

I consent to participate in the project and for my personal data to be used as described.

Place and Date
Participant's Signature
Participant's Name in Block Letters